CLINICAL TRIAL: NCT00592072
Title: Effect of Medium Chain Fatty Acids on Cognitive Function During Acute Hypoglycemia in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK66108b_0505000079; R37DK020495 (NIH); DK20495
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Medium Chain Fatty Acid; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — decanoic acid; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medium chain fatty acid (Octanoic and Decanoic acid) (Experimental)
  Interventions: Dietary Supplement: Medium chain fatty acid (Octanoic and Decanoic acid)
- Splenda (Placebo Control) (Placebo Comparator)
  Interventions: Other: Splenda (Placebo Control)

INTERVENTIONS:
Dietary Supplement: Medium chain fatty acid (Octanoic and Decanoic acid) — Octanoic acid(67%) and Decanoic acid (27%); MCFA 50g total at 25 minute intervals with front loading of 20g then 10g for three administrations.
  Other Names: Medium Chain Triglycerides; Octanoic and Decanoic acid; Fractionated coconut oil
  Arms: Medium chain fatty acid (Octanoic and Decanoic acid)
Other: Splenda (Placebo Control) — Placebo drink will consist of dietary sweetener Splenda mixed in water at a concentration of 1g/100mL. An unsweetened cherry flavor Koolaid mix will be added at a concentration of 0.3g/100mL of the Splenda drink to enhance flavor.
  Arms: Splenda (Placebo Control)

SUMMARY:
At present, there are no therapeutic agents that can minimize severe hypoglycemia (low blood sugar) and its effects on long-term brain function. The aim of this study is to determine whether the human brain is able to use medium chain fatty acids (MCFA) and/or their metabolites as an alternative fuel source during acute hypoglycemia in patients with Type 1 Diabetes Mellitus (T1DM). The hypothesis is that medium chain fatty acids will provide a rapidly absorbed, non-carbohydrate fuel that will improve cognitive performance during episodes of hypoglycemia (low blood sugar.)

DETAILED DESCRIPTION:
Twelve subjects between the ages of 18 years and 55 years who have had Type 1 Diabetes Mellitus for more than five years and have had tight control of their diabetes as determined by screening blood work will be invited to participate. Each study subject will undergo two hypoglycemic clamp studies (a procedure where the blood sugar is closely regulated with intravenous insulin and glucose.) In these hypoglycemic clamp studies, cognitive testing will be performed during 90 minutes of normal blood glucose followed by 90 minutes of hypoglycemia. During the hypoglycemic period, either the MCFA or a placebo will be administered. Each subject will experience both conditions. The order in which the MCFA is given will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus for greater than 5 years (C-peptide negative)
* Age 18-55 years
* Subject is on intensive insulin therapy resulting in a Hemoglobin A1c of less than 7.5%
* History of frequent hypoglycemic events as defined as having at least one blood glucose of less than 60 mg/dl in the last four weeks

Exclusion Criteria:

* History of hypoglycemia induced seizures
* Pregnancy
* Significant baseline anemia (hemoglobin < 11.0g/dl or hematocrit < 33%)
* A history of liver cirrhosis or porto-caval shunt surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MCT Intervention First, Then Placebo: A total of 40 grams of medium-chain triglycerides (derived from coconut oil containing 67% octanoate, 27% decanaote, and 6% other fatty acids) is ingested at 25-min intervals with front loading of 20 grams then 10 grams twice
- Placebo Intervention First, Then MCT Intervention: A total of 40 grams of cherry-flavored water sweetened with sucralose is ingested at 25-min intervals with front loading of 20 grams then 10 grams twice
Period: First Sequence
Arm/Group | MCT Intervention First, Then Placebo | Placebo Intervention First, Then MCT Intervention
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Wash Out Period
Arm/Group | MCT Intervention First, Then Placebo | Placebo Intervention First, Then MCT Intervention
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Second Sequence
Arm/Group | MCT Intervention First, Then Placebo | Placebo Intervention First, Then MCT Intervention
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline number of subjects reflects the number of subjects with baseline data
Groups:
- Overall Number of Subjects: 12 subjects started the study and 10 completed the study, however 11 subjects are reported in the baseline characteristics because one subjects withdrew before baseline data was collected.
Arm/Group | Overall Number of Subjects
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Immediate Verbal Memory
Description: Results of cognitive function in diabetic patients using tests such as digit symbol substitution (a test of memory), tests of everyday attention, telephone book searching and map searching during either administration of medium chain triglyceride oil or a control solution. The goal was to determine whether the human brain is able to use medium-chain fatty acids (MCFA) and /or their metabolites as an alternative fuel source and thus improve brain function during acute hypoglycemia in patients with type 1 diabetes. The lowest score is 0 and the highest score is 25. A higher score is an improvement.
Time Frame: 90 minutes
Population: With the validation span test, a decrease in cognitive performance from euglycemia to hypoglycemia (22+/-2.3 vs 13.4+/-2.5) or a difference of 8.6 has been reported. Using this, a sample size of 12 will provide 80% power to detect a 23% (i.e. 2 unit) attenuation of the effect of hypoglycemia on cognitive performance.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Type 1 Diabetes With MCT Oil: Subjects ingested a drink containing MCT oil prior to euglycemic-hypoglycemic clamp.
- Type 1 Diabetes Without MCT Oil: Subjects ingested a drink without MCT oil prior to euglycemic-hypoglycemic clamp.
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 15.85 (0.66) | 17.36 (13.28)
  Hypoglycemia | 14.97 (1.13) | 13.28 (1.04)

2. Primary Outcome: Delayed Verbal Memory
Description: The highest score is 25 and the lowest score is 0. The higher scored indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 14.82 (1.25) | 15.33 (1.40)
  Hypoglycemia | 14.80 (1.31) | 11.58 (0.71)

3. Primary Outcome: Verbal Memory Recognition
Description: The highest score is 15. The lowest score is 0. Higher scores indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 13.19 (0.53) | 14.27 (0.23)
  Hypoglycemia | 13.29 (0.50) | 12.14 (0.19)

4. Primary Outcome: Digit Span Backward
Description: The highest score is 35. The lowest score is 0. The higher the score indicates an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 0.60 (0.05) | 0.64 (0.05)
  Hypoglycemia | 0.58 (0.05) | 0.54 (0.05)

5. Primary Outcome: Letter/Number Sequencing
Description: The highest score is 21. The lowest score is 0. Higher scores indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 12.04 (0.81) | 11.07 (0.85)
  Hypoglycemia | 10.97 (0.76) | 9.92 (0.71)

6. Primary Outcome: Digit Symbol Coding
Description: The highest score is 133. The lowest score is 0. Higher scores indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 72.50 (5.27) | 74.04 (4.59)
  Hypoglycemia | 74.99 (4.56) | 68.56 (3.54)

7. Primary Outcome: Map Search (2min)
Description: The highest score is 80. The lowest score is 0. Higher scores indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 73.30 (1.70) | 75.04 (1.92)
  Hypoglycemia | 75.11 (1.51) | 74.67 (1.51)

8. Primary Outcome: Map Search (1min)
Description: The highest score is 80. The lowest score is 0. Higher scores indicate an improvement.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
units on a scale
  Euglycemia | 53.11 (4.16) | 50.35 (3.27)
  Hypoglycemia | 48.42 (3.19) | 42.94 (2.31)

9. Primary Outcome: Telephone Search
Description: This is a ratio of how many symbols are found during a certain period of time. The highest ratio is the best result.
Time Frame: 90 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: symbols/ 90 min
Arm/Group | Type 1 Diabetes With MCT Oil | Type 1 Diabetes Without MCT Oil
Number analyzed (Participants) | 10 | 10
symbols/ 90 min
  Euglycemia | 2.86 (0.17) | 3.14 (0.26)
  Hypoglycemia | 3.06 (0.20) | 3.46 (0.34)

ADVERSE EVENTS:
Arm/Group | MCT Intervention | Placebo Intervention
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCT Intervention (N=12) | Placebo Intervention (N=12)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
No technical limitations were seen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes